CLINICAL TRIAL: NCT01538602
Title: Mean Platelet Volume and TXA2 Levels in Patients With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: MPV_PCOS
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; cardiovascular disorders
MeSH Terms: conditions — Polycystic Ovary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- PCOS patients
- Healthy volunteers

SUMMARY:
Polycystic ovary syndrome (PCOS)is closely associated with insulin resistance and hyperinsulinemia as well as with increased incidence in diabetes, hypertension, dyslipidemia and atherosclerosis. Indeed, subjects with PCOS were reported to carry an increased long-term cardiovascular risk, among others. Aiming to correlate the mean platelet volume, the thromboxane A2 level and the PCOS, an observational study was planned. Clinical evaluation of metabolic outcomes in PCOS patients is compared to a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Women fulfilled two out of three diagnostic criteria for PCOS

Exclusion Criteria:

* Pre-existing secondary endocrine disorders
* History of hypertension, diabetes mellitus or cardiovascular disorders
* Pharmacologic treatment in the last 6 months before entering the study.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Volunteers
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Mean platelet volume
Thromboxane A2

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Patologia Ostetrica e Ginecologica, Catania, Italy